CLINICAL TRIAL: NCT05122455
Title: Effects of Edoxaban on Platelet Aggregation in Patients With Stable Coronary Artery Disease
Brief Title: Effects of Edoxaban on Platelet Aggregation
Acronym: Edoxaban
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Jose Carlos Nicolau, Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: SDC 5189/20/218
Record Dates: First submitted 2021-10-19; First posted 2021-11-16 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: SCAD; AMI
Keywords: edoxaban; direct factor Xa inhibitor; stable coronary artery disease; aspirin; clopidogrel; platelet aggregation
MeSH Terms: interventions — Clopidogrel; edoxaban

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-randomized, interventional study of SCAD patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- ASA baseline (Experimental): Patients in chronic use of ASA
  Interventions: Drug: ASA
- ASA + Edoxaban (Experimental): During this intervention phase, eligible patients will sequentially receive ASA 100 mg 1x/day + edoxaban 60 mg 1x/day for a period of 10 ± 2 days.
  Interventions: Drug: ASA; Drug: Edoxaban
- Clopidogrel (Experimental): Subsequently, ASA and edoxaban will be suspended and clopidogrel 75 mg once a day will be administered for 10 ± 2 days (washout period of the ASA).
  Interventions: Drug: Clopidogrel
- Clopidogrel + Edoxaban (Experimental): Subsequently, it will be associated with edoxaban 60 mg once a day to clopidogrel 75 mg once a day for 10 ± 2 days
  Interventions: Drug: Clopidogrel; Drug: Edoxaban
- Edoxaban (Experimental): Finally, only edoxaban 60 mg once a day for 10 ± 2 days will be administered.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: ASA — During the intervention phases, eligible patients will sequentially receive ASA 100 mg 1x/day + edoxaban 60 mg 1x/day for a period of 10 ± 2 days. Subsequently, ASA and edoxaban will be suspended and clopidogrel 75 mg once a day will be administered for 10 ± 2 days (washout period of the ASA). Subsequently, it will be associated with edoxaban 60 mg once a day to clopidogrel 75 mg once a day for 10 ± 2 days and, finally, only edoxaban 60 mg once a day for 10 ± 2 days will be administered. After the end of the interventions, the ASA 100 mg once a day will be restarted.
  Arms: ASA + Edoxaban; ASA baseline
Drug: Clopidogrel — During the intervention phases, eligible patients will sequentially receive ASA 100 mg 1x/day + edoxaban 60 mg 1x/day for a period of 10 ± 2 days. Subsequently, ASA and edoxaban will be suspended and clopidogrel 75 mg once a day will be administered for 10 ± 2 days (washout period of the ASA). Subsequently, it will be associated with edoxaban 60 mg once a day to clopidogrel 75 mg once a day for 10 ± 2 days and, finally, only edoxaban 60 mg once a day for 10 ± 2 days will be administered. After the end of the interventions, the ASA 100 mg once a day will be restarted.
  Arms: Clopidogrel; Clopidogrel + Edoxaban
Drug: Edoxaban — During the intervention phases, eligible patients will sequentially receive ASA 100 mg 1x/day + edoxaban 60 mg 1x/day for a period of 10 ± 2 days. Subsequently, ASA and edoxaban will be suspended and clopidogrel 75 mg once a day will be administered for 10 ± 2 days (washout period of the ASA). Subsequently, it will be associated with edoxaban 60 mg once a day to clopidogrel 75 mg once a day for 10 ± 2 days and, finally, only edoxaban 60 mg once a day for 10 ± 2 days will be administered. After the end of the interventions, the ASA 100 mg once a day will be restarted.
  Arms: ASA + Edoxaban; Clopidogrel + Edoxaban; Edoxaban

SUMMARY:
Rationale: The interaction between nonvitamin K oral anticoagulants (NOACs) and platelet aggregation is complex. The direct activated factor X inhibitors (factor Xa inhibitors) an NOAC antagonizes thrombin generation, one of most important platelet agonist, so that, factor Xa inhibitors has a potential effect in decreasing thrombin-mediated platelet aggregation. On the other hand, patients who experience ACS continue to have a hypercoagulable state for long periods after the index event. The COMPASS trial showed that, in patients with stable coronary artery disease (SCAD), Rivaroxaban (a direct anti-Xa inhibitor) in addition to antiplatelet agent, compared to antiplatelet therapy alone, reduced the composite endpoint of myocardial infarction, stroke and death.

Objective: Analyze the role of edoxaban on platelet aggregation in SCAD patients.

Methods and Results: This is a prospective, non-randomized, interventional study of SCAD patients taking low-dose acetylsalicylic acid (ASA). Subjects initially will receive in the following sequence: ASA 100 mg once daily (QD) plus edoxaban 60 mg QD, clopidogrel 75 mg QD alone, clopidogrel 75 mg QD plus edoxaban 60 mg QD, and edoxaban 60 mg QD alone. Platelet function will be assessed by standard of care technology, at baseline and after each intervention phase, by Multiplate-ADP® (primary endpoint), Multiplate-Aspi® and Multiplate-TRAP®. In addition to immature platelets fraction (% IPF) and count (IPC). Coagulability will be assessed, at baseline and after each intervention phase, by thromboelastogram (TEG) assessment. Specifically, after the phases in which edoxaban will be administered activated factor X (FXa) level and Plasminogen activator inhibitor-1 (PAI-1) will be evaluated in addition to previous. Finally, inflammatory markers will be, at same way, assessed at baseline and after intervention each phase: ultrasensitive C-reactive protein (us-PCR).

Keywords: edoxaban, direct factor Xa inhibitor, stable coronary artery disease, aspirin, clopidogrel, platelet aggregation.

DETAILED DESCRIPTION:
1. Introduction:

Stable coronary artery disease (SCAD) is the leading cause of deaths attributable to cardiovascular disease in the United States. 720,000 new coronary events are expected - defined as the first acute myocardial infarction (AMI) hospitalized or death from SCAD - and approximately 335,000 recurring events per year.

Patients who survive the initial phase of acute coronary syndrome (ACS) remain at risk of cardiac complications: sudden death, (re) infarction or recurrent rest angina, complications related to the development of coronary thrombosis.

The most common cause of coronary thrombosis is plaque rupture followed by plaque erosion. The plaque rupture represents a stimulus for both thrombosis and coagulation, because thrombin activates platelets and converts fibrinogen into fibrin, characteristic of the "white" arterial thrombus. Therefore, the process of arterial thrombus generation involves both platelet aggregation and blood coagulation.

The importance of the coagulation system underlying plaque complications was addressed by Ardissino et al. in the Global Use of Strategies To Open ocluded coronary artteries (GUSTO) IIb, a prospective multicenter cohort study that evaluated the importance of persistently elevated thrombin generation for outcome in 319 consecutive patients with ACS. In this study, the authors concluded that after an episode of ACS, thrombin generation levels were significantly correlated with a worse U-shaped result.

Orbe et al. showed that patients with a previous history of ACS being treated with platelet antiaggregants generated a higher amount of thrombin, earlier and faster, when compared to stable patients. Their results suggest that these patients could benefit from more potent antithrombotic/anticoagulant agents to prevent thrombin activation and generation. Different anticoagulant drugs have been studied for secondary prevention after ACS to reduce mortality and recurrence of ischemic events.

Directly activated X factor inhibitors (factor Xa inhibitors) antagonize thrombin generation. Two representatives of this class (rivaroxaban and apixaban) were evaluated in the context of ACS:

Atlas ACS-2, a phase III trial, was designed to evaluate the effect of low-dose rivaroxaban (2.5-5 mg twice daily), versus placebo in 15,526 patients with recent ACS. The primary outcome composed of cardiovascular death, AMI or stroke was significantly reduced with both doses compared to placebo (8.9% vs. 10.7%, HR 0.84 P = 0.008). Major hemorrhagic events were higher with rivaroxaban in both doses when compared with placebo (2.1% vs. 0.6%, P <0.001); there were fewer fatal hemorrhagic events with the lowest dose of rivaroxaban compared to the highest dose (0.1% vs. 0.4%, respectively, P = 0.04).

APPRAISE-2 was a randomized, double-blind, placebo-controlled phase III study that compared apixaban (5 mg twice daily) with placebo, in addition to standard antiplatelet therapy, in patients with recent ACS. It was discontinued prematurely after recruiting 7,392 patients because major bleeding events were significantly greater in the apixaban group (1.3% apixaban vs. 0.5% control, HR 2.59; P = 0.001) in the absence of a counterbalance reduction in recurrent ischemic events: primary endpoint (cardiovascular death, AMI, or ischemic stroke) 7.5% event rate in the apixaban v group. 7.9% in the placebo group, HR 0.95; P = 0.51.

In patients with SCAD, the phase III COMPASS study involved 27,395 subjects randomized to receive rivaroxaban 2.5 mg twice daily plus aspirin (ASA) 100 mg once daily, rivaroxaban 5 mg twice daily, or ASA 100 mg once a day. The incidence of the primary composite endpoint of cardiac death, stroke, or AMI was significantly lower in the rivaroxaban plus aspirin group compared to the aspirin-only group (4.1 versus 5.4%; HR = 0.76; P <0.001). On the other hand, major bleeding events were significantly higher in the rivaroxaban plus aspirin group compared to the aspirin only group (HR 1.7; P < 0.001), but intracranial and fatal bleeding events were similar in both groups. In patients with an indication for anticoagulation after an ACS episode (e.g. patients with atrial fibrillation), guidelines recommend the use of triple antithrombotic therapy (double antiplatelet in addition to anticoagulant) initially, followed by dual antithrombotic therapy for 1 month to one year, and after 1 year only keep the anticoagulant. However, in cases of very high ischemic risk, especially if there is a low hemorrhagic risk, some choose to keep the antiplatelet drug at the same time and the antiplatelet drug can be maintain.

Therefore, the demonstration of antiplatelet activity in a factor Xa inhibitor would be useful, in order to reinforce its use in isolation after the first year of the acute episode, even in patients with high ischemic risk. It has been shown in vitro that edoxaban, a direct factor Xa inhibitor, is a potent inhibitor of tissue factor-induced platelet aggregation, and its use has increased the antiplatelet effects of clopidogrel and aspirin. Despite this in vitro demonstration, there are no in vivo studies analyzing the action of this drug on platelet reactivity. The present project was designed to provide information on this important issue, analyzing the role of edoxaban on platelet aggregation in patients with SCAD or a history of AMI for more than 12 months.

2.1 Primary objective: To compare platelet aggregability in patients with SCAD using the Multiplate-TRAP® method at the start of ASA use and after 10 ± 2 days of the association of edoxaban and ASA.

2.2 Secondary objective:

Comparison of platelet aggregability in different scenarios:

1.1.1 Measured by Multiplate-ADP®, Multiplate-Aspi® at baseline and after 10 ± 2 days of edoxaban and ASA.

1.1.2 Measured by Multiplate-ADP®, Multiplate-Aspi® and Multiplate-TRAP® before and after 10 ± 2 days of edoxaban and clopidogrel compared to clopidogrel alone; 1.1.3 Measured by Multiplate-ADP®, Multiplate-Aspi® and Multiplate-TRAP® before and after 10 ± 2 days of edoxaban only compared to AAS only; 1.1.4 Measured by Multiplate-ADP®, Multiplate-Aspi® and Multiplate-TRAP® before and after 10 ± 2 days of edoxaban only compared to clopidogrel alone; 1.1.5 Measured by Multiplate-ADP®, Multiplate-Aspi® and Multiplate-TRAP® before and after 10 ± 2 days of edoxaban plus clopidogrel compared to 10 ± 2 days of edoxaban and AAS.

2.3 Other secondary goals: 1.1.6 Dosage of the following parameters:

1. Total immature platelets (IPC) and fractions (%IPF), and inflammatory markers: ultrasensitive CRP after each intervention phase.
2. Thromboelastography (TEG) after each intervention phase.
3. Dosing of plasminogen activator inhibitor type 1 (PAI-1) and factor Xa activity after each intervention phase in which edoxaban is administered.
4. Analyze the primary objective of the study in the following subgroups:

   * Gender (male/female);
   * Diabetes (presence or not);
   * Current or not smoking;
   * Elderly (≥ 65 years old) and non-elderly.

     3. Methods: 3.1. Study design: Prospective, open, intervention, non-randomized study that will be conducted at Heart Institute (InCor) HCFMUSP.

After signing the free and informed consent form , the patient will undergo a physical examination and be classified by the HAS-BLED according to the risk of bleeding; then, blood samples will be collected for safety assessment (complete blood count, coagulation, kidney and liver function tests).

Eligible patients for the study will be evaluated at five more visits in addition to the screening visit. In four of the remaining visits there will be different interventions (first visit, second visit, third visit and fourth visit).

The following laboratory tests will be performed at the beginning and after each intervention phase: Multiplate-ADP®, Multiplate-Aspi®, Multiplate-TRAP®, IPF and IPC; Ultrasensitive PCR and TEG. Specifically, after the phases in which edoxaban will be administered, FXa and PAI-1 level activity will be further evaluated.

3.2. Study procedures:

During the intervention phases, eligible patients will sequentially receive ASA 100 mg 1x/day + edoxaban 60 mg 1x/day for a period of 10 ± 2 days. Subsequently, ASA and edoxaban will be suspended and clopidogrel 75 mg once a day will be administered for 10 ± 2 days (washout period of the ASA). Subsequently, it will be associated with edoxaban 60 mg once a day to clopidogrel 75 mg once a day for 10 ± 2 days and, finally, only edoxaban 60 mg once a day for 10 ± 2 days will be administered. After the end of the interventions, the ASA 100 mg once a day will be restarted. All study medications and procedures will be fully paid for by those responsible for the study, without any burden to the Unified Health System or to Supplementary Health.

Criteria for stopping current medication:

The study drug should be discontinued in the event of major bleeding, defined by the presence of at least one of the following criteria: fall in hemoglobin level greater than or equal to 2.0g/dL or transfusion of two or more units of packed red blood cells; bleeding from a critical site or organ such as intracranial, intraspinal, intraocular, pericardial, intraarticular, intramuscular with compartment syndrome, retroperitoneal; or fatal hemorrhage.

Bleeding that does not meet the criteria for major bleeding, but that has been associated with a medical intervention, an unscheduled contact (visit) with a physician, or associated with discomfort for the subject, such as pain or impairment of activities of daily living will be considered clinically relevant, but not severe bleeding.

3.3. Selection: The patients included will be selected from the outpatient clinics of the Heart Institute (InCor) HCFMUSP and from the database of the Thematic project "Platelet aggregation and antiaggregation in patients with coronary artery disease" (SDC 4086 /14/066; FAPESP 2014/01021-4) of the InCor Acute Coronary Disease Unit.

3.4. Inclusion criteria:

1. Patients aged between 18 and 75 years
2. Confirmed diagnosis of CAD using ASA 100 mg once a day. The following will be considered for SCAD diagnosis: previous history of type 1 AMI (at least one year ago), according to the fourth universal definition of myocardial infarction and/or coronary angioplasty and/or coronary artery bypass graft surgery myocardium and/or coronary angiography showing at least 50% obstruction in one of the main epicardial vessels.
3. Agreement to sign the free and informed consent form.

3.5. Exclusion criteria:

* Clinically active bleeding or clinically significant bleeding in the last year.
* Peptic ulcer active in the last 60 days
* Previous history of high gastrointestinal bleeding
* Hemoglobin <10 g / dl at randomization;
* Platelets <100,000 or >500,000 µ/L
* Need for lumbar puncture
* Atrial fibrillation
* Metal valve prosthesis
* Percutaneous coronary intervention (PCI) in the last 3 months with conventional stent and in the last 6 months with drug-eluting stent.
* Surgical myocardial revascularization (CABG) in the last 90 days
* Percutaneous coronary intervention (PCI) or surgical myocardial revascularization (CABG) planned within the next 60 days;
* Previous hemorrhagic stroke;
* Moderate or severe liver failure associated with coagulation disorders (Child-Pugh B or C)
* Hypersensitivity to edoxaban or formula components;
* Pregnant women or women of childbearing potential;
* Chronic kidney disease: glomerular filtration rate estimated at <50 mL/min/1.73m², calculated using the Cockcroft-Gault equation;
* Current or last 30 days use of anticoagulant or antiplatelet therapy, except ASA;
* Weight <60 kg;
* HAS-BLED score ≥ 3 points;
* Concomitant use of P-glycoprotein inhibitors such as azithromycin, clarithromycin, erythromycin, itraconazole, ketoconazole, verapamil, quinidine, except amiodarone;
* Concomitant use of P-glycoprotein inducers, such as Rifampicin;
* Known abuse of alcohol, drugs, or medications in the 12 months prior to consent for this study;
* Cancer therapy 5 years prior to consent for this study;
* Medicines that will further increase the risk of bleeding (such as nonsteroidal anti-inflammatory drugs).
* Participation in another study within 30 days of signing the consent form.

3.6. Procedures

Blood samples:

All blood samples will be collected between 8:00 am and 12:00 pm (2 to 4 hours after the last drug ingestion), after 30 minutes of rest, by antecubital venipuncture with a 21-gauge needle. Within 2 hours after collection, platelet function tests (Multiplate®) will be performed. The other samples will be centrifuged at 3,000 rpm, stored in aliquots and subsequently frozen at -80 degrees Celsius for further analysis by enzyme immunoassay (ELISA).

Description of laboratory tests:

1. Multiple electrode aggregometry - MEA (Multiplate® from Roche): a volume of 3.0 ml of blood will be collected in a hirudin tube, 300 µL of this sample is diluted with 300 µL of 0.9% NaCl and incubated in a test cuvette at 37°C for 3 minutes. Then, as recommended by the manufacturer, platelet aggregation will be induced by the addition of arachidonic acid (ASPItest), ADP (ADPtest) or TRAP-6 (TRAPtest). The platelet aggregation response will be continuously recorded for 6 minutes. The increase in impedance due to the fixation of platelets to the electrodes is detected for each sensor unit separately and transformed into aggregation units (AU) which are plotted. Approximately 8 AU corresponds to 1 Ohm. Aggregation measured with Multiplate® is quantified as AU and area under the curve (AUC) of aggregation units (AU * min). Multiplate® displays and documents aggregation tracings providing a qualitative assessment of platelet function;
2. PCRus: will be determined by the IMMULITE automated analyzer (Immulite, DPC medLAB, Los Angeles, USA).
3. PAI-1 inhibits the serine protease urokinase (uPA) and tissue plasminogen activator (tPA), resulting in the inhibition of fibrinolysis. The elevation of plasma PAI-1 has been described as a prothrombotic factor in arterial and venous thromboembolic disorders. Furthermore, high levels of PAI-1 are associated with an increased incidence of acute coronary syndromes. The determination of plasma PAI-1 will be performed by ELISA.
4. ROTEM: The viscoelastic properties of the clot, such as clot formation (clotting time and clot formation time), clot strength (maximum clot firmness), alpha angle and clot lysis, will be determined using the ROTEM delta device (Instrumentation Laboratory, Bedford, MA, USA).
5. Anti-XA: The Liquid Anti-Xa chromogenic method will be performed with specific calibrators and controls for edoxaban, manufacturer Stago (Diagnostica Stago, France) in automated coagulation equipment STA-R® and STA Compact® (Diagnostica Stago, France). STA® Liquid Anti-Xa are intended for the quantitative determination in plasma of edoxaban, measuring its direct anti-Xa activity in a competitiveness study.

   Edoxaban levels are given in ng/mL. The detection limit on the STA-R® and STA Compact® is 20 ng/mL and the linearity range extends up to 400 ng/mL. The test will be performed on platelet poor plasma (PPP).

   4. Sample size

   Previous publications analyzing platelet aggregation in patients with CAD by Multiplate-TRAP® (Roche) showed a mean platelet reactivity of 102 ± 26 AUC. Assuming that the standard deviation of the difference is the same standard deviation as the mean, and a 20% decrease in platelet aggregability after the use of edoxaban, an alpha error of 0.01 two-tailed (considering the multiplicity adjustment by Bonferroni - see below) and a power of 95%, a sample size of 57 patients was obtained. Based on these calculations and considering possible losses to follow-up (approximately 20%), we propose a sample of 70 patients to be analyzed in this study.

   5. Statistical analysis The results will be presented as number and percentage (categorical variables); continuous variables will be presented as means ± SD (Gaussian distribution) or medians and interquartile values (non-Gaussian distribution). Due to the paired design, the interest groups will not be independent from each other. Because of this, comparisons between them in relation to continuous variables will be made using the Student t test for paired samples, for variables with normal distribution, or the Wilcoxon signed rank test, for non-Gaussian distribution variables. Due to the multiplicity of hypotheses (5 in total), the sample size calculation has already been adjusted by Bonferroni, leading to an overall type 1 error of 5%. Therefore, for each individual comparison (edoxaban + aspirin versus aspirin, edoxaban + clopidogrel versus clopidogrel, etc.), a p<0.01 will be considered statistically significant. Regarding the tests, the multiplicity adjustment will take into account the Multiplate-TRAP®, while Multiplate-ADP® and Multiplate-Aspi® will be considered exploratory.

   6. Ethical issues: This protocol is in accordance with the recommendations contained in the Declaration of Helsinki and was approved, together with the Informed Consent Form (attached), by the Scientific Committee of InCor and by the Research Ethics Committee of HC/FMUSP (CAAE:43768921.6.0000.0068).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years
* Confirmed diagnosis of CAD using ASA 100 mg once a day. The following will be considered for CAD diagnosis: previous history of type 1 AMI (at least one year ago), according to the fourth universal definition of myocardial infarction (Thygesen, Alpert et al. 2018) and/or coronary angioplasty and/or coronary artery bypass graft surgery myocardium and/or coronary angiography showing at least 50% obstruction in one of the main epicardial vessels.
* Agreement to sign the free and informed consent form.

Exclusion Criteria:

* Clinically active bleeding or clinically significant bleeding in the last year.
* Peptic ulcer active in the last 60 days
* Previous history of high gastrointestinal bleeding
* Hemoglobin <10 g / dl at randomization;
* Platelets <100,000 or >500,000 µ/L
* Need for lumbar puncture
* Atrial fibrillation
* Metal valve prosthesis
* Percutaneous coronary intervention (PCI) in the last 3 months with conventional stent and in the last 6 months with drug-eluting stent.
* Surgical myocardial revascularization (CABG) in the last 90 days
* Percutaneous coronary intervention (PCI) or surgical myocardial revascularization (CABG) planned within the next 60 days;
* Previous hemorrhagic stroke;
* Moderate or severe liver failure associated with coagulation disorders (Child-Pugh B or C)
* Hypersensitivity to edoxaban or formula components;
* Pregnant women or women of childbearing potential;
* Chronic kidney disease: glomerular filtration rate estimated at <50 mL/min/1.73m², calculated using the Cockcroft-Gault equation;
* Current or last 30 days use of anticoagulant or antiplatelet therapy, except ASA;
* Weight <60 kg;
* HAS-BLED score ≥ 3 points;
* Concomitant use of P-glycoprotein inhibitors such as azithromycin, clarithromycin, erythromycin, itraconazole, ketoconazole, verapamil, quinidine, except amiodarone;
* Concomitant use of P-glycoprotein inducers, such as Rifampicin;
* Known abuse of alcohol, drugs, or medications in the 12 months prior to consent for this study;
* Cancer therapy 5 years prior to consent for this study;
* Medicines that will further increase the risk of bleeding (such as nonsteroidal anti-inflammatory drugs).
* Participation in another study within 30 days of signing the consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Main objective: | 24 months
  To compare platelet aggregability in patients with CAD using the Multiplate-TRAP® method at the start of ASA use and after 10 ± 2 days of the association of edoxaban and ASA.

SECONDARY OUTCOMES:
Platelet reactivity after edoxaban plus ASA vs ASA | 24 months
  To compare of platelet aggregability measured by Multiplate-ADP®, Multiplate-Aspi® at baseline and after 10 ± 2 days of edoxaban and ASA.
Platelet reactivity after edoxaban plus Clopidogrel vs Clopidogrel | 24 months
  To compare of platelet aggregability measured by Multiplate-ADP®, Multiplate-Aspi® and Multiplate-TRAP® before and after 10 ± 2 days of edoxaban and clopidogrel compared to clopidogrel alone;
Platelet reactivity after edoxaban vs after ASA | 24 months
  To compare of platelet aggregability measured by Multiplate-ADP®, Multiplate-Aspi® and Multiplate-TRAP® before and after 10 ± 2 days of edoxaban only compared to ASA only;
Platelet reactivity after edoxaban vs after Clopidogrel | 24 months
  To compare of platelet aggregability measured Multiplate-ADP®, Multiplate-Aspi® and Multiplate-TRAP® before and after 10 ± 2 days of edoxaban only compared to clopidogrel alone;
Platelet reactivity after edoxaban plus ASA vs after edoxaban plus Clopidogrel | 24 months
  To compare of platelet aggregability measured Multiplate-ADP®, Multiplate-Aspi® and Multiplate-TRAP® before and after 10 ± 2 days of edoxaban plus clopidogrel compared to 10 ± 2 days of edoxaban and AAS.

OTHER OUTCOMES:
Other secondary goals | 24 months
  1. Total immature platelets (IPC) and fractions (%IPF), and inflammatory markers: ultrasensitive CRP after each intervention phase.
  2. Thromboelastography (TEG) after each intervention phase.
  3. Dosing of plasminogen activator inhibitor type 1 (PAI-1) and factor Xa activity after each intervention phase in which edoxaban is administered.
  4. Analyze the primary objective of the study in the following subgroups:
     * Gender (male/female);
     * Diabetes (presence or not);
     * Current or not smoking;
     * Elderly (≥ 65 years old) and non-elderly.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coracao (InCor), Hospital das Clinicas HCFMUSP, Faculdade de Medicina, Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Alexander JH, Lopes RD, James S, Kilaru R, He Y, Mohan P, Bhatt DL, Goodman S, Verheugt FW, Flather M, Huber K, Liaw D, Husted SE, Lopez-Sendon J, De Caterina R, Jansky P, Darius H, Vinereanu D, Cornel JH, Cools F, Atar D, Leiva-Pons JL, Keltai M, Ogawa H, Pais P, Parkhomenko A, Ruzyllo W, Diaz R, White H, Ruda M, Geraldes M, Lawrence J, Harrington RA, Wallentin L; APPRAISE-2 Investigators. Apixaban with antiplatelet therapy after acute coronary syndrome. N Engl J Med. 2011 Aug 25;365(8):699-708. doi: 10.1056/NEJMoa1105819. Epub 2011 Jul 24. PMID 21780946
- [Background] Angiolillo DJ, Bhatt DL, Cannon CP, Eikelboom JW, Gibson CM, Goodman SG, Granger CB, Holmes DR, Lopes RD, Mehran R, Moliterno DJ, Price MJ, Saw J, Tanguay JF, Faxon DP. Antithrombotic Therapy in Patients With Atrial Fibrillation Treated With Oral Anticoagulation Undergoing Percutaneous Coronary Intervention: A North American Perspective: 2021 Update. Circulation. 2021 Feb 9;143(6):583-596. doi: 10.1161/CIRCULATIONAHA.120.050438. Epub 2021 Feb 8. PMID 33555916
- [Background] Arantes FBB, Menezes FR, Franci A, Barbosa CJDG, Dalcoquio TF, Nakashima CAK, Baracioli LM, Furtado RHM, Nomelini QSS, Ramires JAF, Kalil Filho R, Nicolau JC. Influence of Direct Thrombin Inhibitor and Low Molecular Weight Heparin on Platelet Function in Patients with Coronary Artery Disease: A Prospective Interventional Trial. Adv Ther. 2020 Jan;37(1):420-430. doi: 10.1007/s12325-019-01153-8. Epub 2019 Nov 22. PMID 31758517
- [Background] Ardissino D, Merlini PA, Bauer KA, Galvani M, Ottani F, Franchi F, Bertocchi F, Rosenberg RD, Mannucci PM. Coagulation activation and long-term outcome in acute coronary syndromes. Blood. 2003 Oct 15;102(8):2731-5. doi: 10.1182/blood-2002-03-0954. Epub 2003 Jul 3. PMID 12843003
- [Background] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Background] Connolly SJ, Eikelboom JW, Bosch J, Dagenais G, Dyal L, Lanas F, Metsarinne K, O'Donnell M, Dans AL, Ha JW, Parkhomenko AN, Avezum AA, Lonn E, Lisheng L, Torp-Pedersen C, Widimsky P, Maggioni AP, Felix C, Keltai K, Hori M, Yusoff K, Guzik TJ, Bhatt DL, Branch KRH, Cook Bruns N, Berkowitz SD, Anand SS, Varigos JD, Fox KAA, Yusuf S; COMPASS investigators. Rivaroxaban with or without aspirin in patients with stable coronary artery disease: an international, randomised, double-blind, placebo-controlled trial. Lancet. 2018 Jan 20;391(10117):205-218. doi: 10.1016/S0140-6736(17)32458-3. Epub 2017 Nov 10. PMID 29132879
- [Background] Freeman MR, Williams AE, Chisholm RJ, Armstrong PW. Intracoronary thrombus and complex morphology in unstable angina. Relation to timing of angiography and in-hospital cardiac events. Circulation. 1989 Jul;80(1):17-23. doi: 10.1161/01.cir.80.1.17. PMID 2736749
- [Background] Furugohri T, Isobe K, Honda Y, Kamisato-Matsumoto C, Sugiyama N, Nagahara T, Morishima Y, Shibano T. DU-176b, a potent and orally active factor Xa inhibitor: in vitro and in vivo pharmacological profiles. J Thromb Haemost. 2008 Sep;6(9):1542-9. doi: 10.1111/j.1538-7836.2008.03064.x. Epub 2008 Jul 4. PMID 18624979
- [Background] Gibson CM, Mega JL, Burton P, Goto S, Verheugt F, Bode C, Plotnikov A, Sun X, Cook-Bruns N, Braunwald E. Rationale and design of the Anti-Xa therapy to lower cardiovascular events in addition to standard therapy in subjects with acute coronary syndrome-thrombolysis in myocardial infarction 51 (ATLAS-ACS 2 TIMI 51) trial: a randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of rivaroxaban in subjects with acute coronary syndrome. Am Heart J. 2011 May;161(5):815-821.e6. doi: 10.1016/j.ahj.2011.01.026. PMID 21570509
- [Background] Honda Y, Kamisato C, Morishima Y. Edoxaban, a direct factor Xa inhibitor, suppresses tissue-factor induced human platelet aggregation and clot-bound factor Xa in vitro: Comparison with an antithrombin-dependent factor Xa inhibitor, fondaparinux. Thromb Res. 2016 May;141:17-21. doi: 10.1016/j.thromres.2016.02.028. Epub 2016 Feb 26. PMID 26962981
- [Background] Honda Y, Kamisato C, Morishima Y. Prevention of arterial thrombosis by edoxaban, an oral factor Xa inhibitor in rats: monotherapy and in combination with antiplatelet agents. Eur J Pharmacol. 2016 Sep 5;786:246-252. doi: 10.1016/j.ejphar.2016.06.011. Epub 2016 Jun 7. PMID 27288116
- [Background] Huber K, Christ G, Wojta J, Gulba D. Plasminogen activator inhibitor type-1 in cardiovascular disease. Status report 2001. Thromb Res. 2001 Sep 30;103 Suppl 1:S7-19. doi: 10.1016/s0049-3848(01)00293-6. PMID 11567664
- [Background] Khalil P, Kabbach G. Direct Oral Anticoagulants in Addition to Antiplatelet Therapy for Secondary Prevention after Acute Coronary Syndromes: a Review. Curr Cardiol Rep. 2019 Jan 28;21(1):5. doi: 10.1007/s11886-019-1088-x. PMID 30689068
- [Background] Lippi G, Franchini M, Targher G. Arterial thrombus formation in cardiovascular disease. Nat Rev Cardiol. 2011 Jul 5;8(9):502-12. doi: 10.1038/nrcardio.2011.91. PMID 21727917
- [Background] Orbe J, Zudaire M, Serrano R, Coma-Canella I, Martinez de Sizarrondo S, Rodriguez JA, Paramo JA. Increased thrombin generation after acute versus chronic coronary disease as assessed by the thrombin generation test. Thromb Haemost. 2008 Feb;99(2):382-7. doi: 10.1160/TH07-07-0443. PMID 18278189
- [Background] Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest. 2010 Nov;138(5):1093-100. doi: 10.1378/chest.10-0134. Epub 2010 Mar 18. PMID 20299623
- [Background] Sibbing D, Braun S, Jawansky S, Vogt W, Mehilli J, Schomig A, Kastrati A, von Beckerath N. Assessment of ADP-induced platelet aggregation with light transmission aggregometry and multiple electrode platelet aggregometry before and after clopidogrel treatment. Thromb Haemost. 2008 Jan;99(1):121-6. doi: 10.1160/TH07-07-0478. PMID 18217143
- [Background] Sibbing D, Aradi D, Alexopoulos D, Ten Berg J, Bhatt DL, Bonello L, Collet JP, Cuisset T, Franchi F, Gross L, Gurbel P, Jeong YH, Mehran R, Moliterno DJ, Neumann FJ, Pereira NL, Price MJ, Sabatine MS, So DYF, Stone GW, Storey RF, Tantry U, Trenk D, Valgimigli M, Waksman R, Angiolillo DJ. Updated Expert Consensus Statement on Platelet Function and Genetic Testing for Guiding P2Y12 Receptor Inhibitor Treatment in Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2019 Aug 26;12(16):1521-1537. doi: 10.1016/j.jcin.2019.03.034. Epub 2019 Jun 12. PMID 31202949
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Hokusai-VTE Investigators; Buller HR, Decousus H, Grosso MA, Mercuri M, Middeldorp S, Prins MH, Raskob GE, Schellong SM, Schwocho L, Segers A, Shi M, Verhamme P, Wells P. Edoxaban versus warfarin for the treatment of symptomatic venous thromboembolism. N Engl J Med. 2013 Oct 10;369(15):1406-15. doi: 10.1056/NEJMoa1306638. Epub 2013 Aug 31. PMID 23991658
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Virmani R, Burke AP, Farb A, Kolodgie FD. Pathology of the vulnerable plaque. J Am Coll Cardiol. 2006 Apr 18;47(8 Suppl):C13-8. doi: 10.1016/j.jacc.2005.10.065. PMID 16631505
- [Background] von Pape KW, Dzijan-Horn M, Bohner J, Spannagl M, Weisser H, Calatzis A. [Control of aspirin effect in chronic cardiovascular patients using two whole blood platelet function assays. PFA-100 and Multiplate]. Hamostaseologie. 2007 Aug;27(3):155-60; quiz 161-2. doi: 10.1007/978-3-540-36715-4_49. German. PMID 17694222
- [Background] Wurtz M, Hvas AM, Christensen KH, Rubak P, Kristensen SD, Grove EL. Rapid evaluation of platelet function using the Multiplate(R) Analyzer. Platelets. 2014;25(8):628-33. doi: 10.3109/09537104.2013.849804. Epub 2013 Nov 18. PMID 24246241